CLINICAL TRIAL: NCT02103660
Title: A Randomized Clinical Trial on the Effects of Progestin-based Contraception in the Genital Tract of HIV-infected and Uninfected Women
Brief Title: Clinical Trial on the Effects of Progestin-based Contraception in the Genital Tract of HIV-infected and Uninfected Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH); Bill and Melinda Gates Foundation (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CDC-NCCDPHP-6512; 1K01TW009657-01 (NIH); U48DP001944 (NIH); SIP 09-022 (Other Grant/Funding Number: CDC); UNCPM 1303 (Other: University of North Carolina)
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: HIV; Contraception
Keywords: contraceptive implant; Depo-Medroxyprogesterone Acetate; Hormonal Contraception; progestin
MeSH Terms: interventions — Medroxyprogesterone Acetate; N,N-dimethyl-4-anisidine; Contraceptive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Depo-Medroxyprogesterone Acetate (Active Comparator): Half of women will be randomized to receive Depo-Medroxyprogesterone Acetate injections every 13 weeks
  Interventions: Drug: Depo-Medroxyprogesterone Acetate
- Progestin Implant (Jadelle) (Active Comparator): Half of women will be randomized to receive progestin implant.
  Interventions: Drug: Progestin Contraceptive (Jadelle)

INTERVENTIONS:
Drug: Depo-Medroxyprogesterone Acetate — 150 mg Depo-Medroxyprogesterone Acetate administered every 13 weeks
  Other Names: Depo provera; DMPA; injectable contraception
  Arms: Depo-Medroxyprogesterone Acetate
Drug: Progestin Contraceptive (Jadelle) — 2 implants containing 75 mg of levonorgestrel will be implanted and will last for up to 5 years
  Other Names: Jadelle; Contraceptive Implant
  Arms: Progestin Implant (Jadelle)

SUMMARY:
The purpose of this study is to determine the acceptability of randomization to contraceptive options and estimate the effect of progestin contraception on HIV genital shedding and inflammatory/immune perturbations in women who may or may not be on antiretroviral therapy, as well as in HIV-uninfected women controls. It is hypothesized that progestin-containing contraception will lead to inflammatory changes that may affect the local immune activity, influencing HIV acquisition or transmissibility risk.

DETAILED DESCRIPTION:
Hormonal contraception is a central component in the prevention of unintended pregnancy; however there are concerns that certain methods may increase the risk of heterosexual HIV acquisition and transmission. Some studies, but not others, have suggested a link between hormonal contraceptive use and enhanced HIV-susceptibility, more rapid HIV disease progression, and increased transmissibility to partners. Hormonal contraception modifies the genital mucosa in several ways, and the interactions of the endocrine and immune system are complex but incompletely understood. In some cross-sectional studies, hormonal contraceptives appear to be associated with increased shedding of HIV DNA, but not RNA, in the genital tract, and the significance of these findings for HIV transmissibility are unclear. Very few studies have examined genital HIV shedding prospectively before and after initiation of contraception. The effects of hormonal contraception in the setting of antiretroviral therapy (ART) are also unknown.

Hormonal contraception, particularly injectable DMPA, is widely used in many parts of the world, including settings with high HIV prevalence. It is important that the effects of hormonal contraception on HIV acquisition and HIV shedding and subsequent transmissibility be determined. The effect of progestin contraceptive implants, such as the levonorgestrel rod implant (LNG implant), on HIV shedding is unknown, and it will be of interest to evaluate it compared with the injectable progestin (DMPA), given their different kinetics of hormone release, differences in progestin type, and the high efficacy of both methods.

We propose a pilot study among 100 HIV-infected women and 30 uninfected women in Lilongwe, Malawi randomized to either DMPA or LNG implant to: 1) assess the effect and compare the impact of type of progestin-containing contraception (injectable versus implant) on HIV viral shedding in the genital tract of HIV+ women, 2) assess the effect and compare the impact of type of progestin-containing contraception (injectable versus implant) on inflammatory/immune markers in the genital tract of both HIV+ and HIV- women, and 3) assess the interaction of progestin-based hormonal contraception and ART by examining: i. contraceptive efficacy (measured by systemic hormone levels and pregnancy rate during follow-up), and ii. ART efficacy (by drug concentrations in blood and genital tract and HIV viral load response in the plasma in women on ART).

An overall study aim is to determine the feasibility and need for a larger study of determinants of HIV transmissibility and acquisition in this population.

The study would take place at Bwaila Maternity Hospital, which was the site of the CDC-sponsored Breastfeeding, Antiretrovirals, and Nutrition (BAN) clinical trial, a partner project with this study. Women attending the clinics at Bwaila (a large proportion of whom participated in the BAN study) who desire to start hormonal contraception will be informed of the new study and counseled on the progestin-based contraceptives that are available within the study. BAN women will be specifically targeted for recruitment through radio messages. Eligible women who provide informed consent and agree to randomization to either DMPA or the LNG implant will be enrolled. HIV-infected women may be on ART or they may be pre-ART.

To address the primary outcomes of HIV shedding and mucosal immune activation, we will quantify genital tract HIV RNA and inflammatory/immune markers at two time points before and four time points after randomization of the 100 HIV-infected and 30 HIV-uninfected women to DMPA or LNG-implant. The two time points prior to randomization will occur within the prior menstrual cycle, so that one visit occurs in the follicular phase and the other occurs in the luteal phase of the cycle. Assessments after initiation of contraception will occur on days 3, 30, 90, and 6 months. Antiretroviral levels in the blood and genital tract will also be assessed at these time points.

Based on recent evidence suggesting that the LNG implant may have decreased contraceptive efficacy when used in combination with the antiretroviral efavirenz, study follow-up will be extended to include visits at about 9, 12, 15, 18, 21, 24, 27, 30, and 33 months after initiation of contraception for a total of 6 additional visits per participant. Not all participants will start the study extension at the same time point, so the 6 additional visits can span from about 9 months to 24 months after contraceptive initiation to about 18 months to 33 months after contraceptive initiation. Assessments at these visits will address the outcomes of contraceptive and ART efficacy and HIV shedding.

To analyze the effects of progestin contraception on HIV shedding, as well as the effect of each contraceptive type, HIV-infected women on progestin-based contraception will be compared within each study arm (before and after initiation of contraception), as well as between the two contraceptive arms. Antiretroviral use will be evaluated for an independent effect on HIV shedding and also to determine if it modifies the effect of menstrual cycle or progestin contraception on HIV shedding. To analyze the effects of progestin contraception on genital inflammatory/immune markers, both HIV-infected and HIV-uninfected women on progestin-based contraception will be compared separately and combined, with HIV status treated as a potential effect modifier, within each study arm (before and after initiation of contraception), as well as between the two contraceptive arms. This study will provide information on acceptability of randomization to contraceptive options, overall study retention, and estimates of the effect of progestin contraception on HIV genital shedding and inflammatory/immune perturbations in women who may or may not be on antiretroviral therapy, as well as in HIV-uninfected women controls. This information will be instrumental in determining the need for and feasibility of a larger study to address these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Known HIV status, as documented by at least 2 concordant rapid tests (Determine and Uni-Gold, respectively). If the 2 rapid tests are discordant, then a confirmatory test will be done via Western blot.
* Female, pre-menopausal, age 18 to 45 years
* At least 2 regular, monthly cycles (~21-35 days) in the 3 months preceding study enrollment.
* If on hormonal or intrauterine contraception in the past, they must have been off for at least 6 months. If they were previously using DMPA, their last -injection must have been ≥6 months ago.
* If recently pregnant, they must be at least 6 months postpartum
* Able and willing to provide informed consent
* Be otherwise a good candidate for study participation based on assessment by investigator or designee
* Interested in initiating a family planning method, specifically depot medroxyprogesterone acetate (DMPA) or the LNG implant (Jadelle)
* Willing to be randomized to receive either DMPA or LNG implant (Jadelle)
* Willing to wait 4-6 weeks after enrollment to receive this method and to use non-hormonal and non-intrauterine methods (such as abstinence or condoms) consistently during this period

Exclusion Criteria:

* Pregnancy (by clinical history or a positive urine pregnancy test at screening)
* Women currently using any hormonal contraceptive method
* Desire pregnancy within next 12 months
* Untreated visible genital ulcers or lesions on initial pelvic examination
* Known or suspected genital tract cancer (by clinical history or noted during initial pelvic examination).
* Contraindications to DMPA or LNG implant per the WHO medical eligibility114 criteria or judgment of clinician (contraindications include lactation within first 6 weeks postpartum, acute deep venous thrombosis or pulmonary embolism, lupus, migraine with aura, unexplained vaginal bleeding, current or history of breast cancer, severe cirrhosis, liver tumors, history of stroke, current or history of ischemic heart disease).
* Acute HIV infection (as documented by a known negative HIV test 6 months or less prior to screening).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2014-04-08 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
HIV viral load in the genital tract of HIV-infected women before and after initiation of progestin-containing contraception | 6 months post randomization; 24 months to 33 months post randomization
  Genital HIV viral load at each study visit will be modeled longitudinally as a continuous outcome using a generalized estimating equation (GEE) model. The model will include a covariate indicating whether the measurement was taken before or after receiving the contraceptive method, and the null hypothesis will be tested using a z-test on this covariate.
HIV viral load in the genital tract of HIV-infected women by contraceptive type | 6 months post randomization;24 months to 33 months post randomization
  Genital HIV viral load at each study visit will be modeled longitudinally as a continuous outcome using a generalized estimating equation (GEE) model. The model will include a covariate for contraception arm, and the null hypothesis will be tested using a z-test on this covariate.

SECONDARY OUTCOMES:
Impact of the type of progestin-containing contraception (injectable versus implant) on inflammatory/immune markers in the genital tract women. | 6 months post randomization
  A series of paired t-tests or Wilcoxon signed-rank tests, with Bonferonni correction, will be used for the within-subject assessments of all the immune markers, before and after contraceptive initiation. The baseline value will be the mean of the follicular and luteal phase values, and it will be compared to the value for each study time point after contraceptive initiation. Comparisons will be performed between subjects in the LNG-implant and DMPA arms.
Contraceptive efficacy in HIV-infected women | 6 months post randomization; 24 months to 33 months post randomization
  Contraceptive efficacy will be measured by the occurrence of any pregnancies and compared by antiretroviral status
Interaction of progestin-based hormonal contraception and antiretroviral therapy | 6 months post randomization;24 months to 33 months post randomization
  Plasma and female genital tract ARV drug concentrations will be expressed as geometric mean with corresponding 95% confidence interval. Correlation between genital tract viral shedding, plasma and genital tract ARV concentrations and hormonal contraception will be assessed with longitudinal models using GEE. Outcomes will be compared between the DMPA and the implant users evaluating the contraceptive method as an effect modifier for HIV shedding or ART concentrations within the longitudinal models.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Tang, MD, MSCR, Study Chair — University of North Carolina; Lameck Chinula, MD, Study Chair — UNC-Project Lilongwe; Athena P Kourtis, MD, PhD, MPH, Study Chair — Centers for Disease Control and Prevention
Locations (1):
- UNC-Project Lilongwe, Lilongwe, Malawi

REFERENCES:
- [Derived] Haddad LB, Tang JH, Davis NL, Kourtis AP, Chinula L, Msika A, Tegha G, Hosseinipour MC, Nelson JAE, Hobbs MM, Gajer P, Ravel J, De Paris K. Influence of Hormonal Contraceptive Use and HIV on Cervicovaginal Cytokines and Microbiota in Malawi. mSphere. 2023 Feb 21;8(1):e0058522. doi: 10.1128/msphere.00585-22. Epub 2023 Jan 9. PMID 36622252
- [Derived] Zia Y, Tang JH, Chinula L, Tegha G, Stanczyk FZ, Kourtis AP. Medroxyprogesterone acetate concentrations among HIV-infected depot-medroxyprogesterone acetate users receiving antiretroviral therapy in Lilongwe, Malawi. Contraception. 2019 Nov;100(5):402-405. doi: 10.1016/j.contraception.2019.07.144. Epub 2019 Jul 30. PMID 31374188
- [Derived] Chinula L, Nelson JAE, Wiener J, Tang JH, Hurst S, Tegha G, Msika A, Ellington S, Hosseinipour MC, Mataya R, Haddad LB, Kourtis AP. Effect of the depot medroxyprogesterone acetate injectable and levonorgestrel implant on HIV genital shedding: a randomized trial. Contraception. 2018 Sep;98(3):193-198. doi: 10.1016/j.contraception.2018.05.001. Epub 2018 May 8. PMID 29746813